CLINICAL TRIAL: NCT02356887
Title: Measurement of Flow in Internal Jugular Vein in the Sitting Position: an Ultrasound Study on Healthy Volunteers
Brief Title: Internal Jugular Vein Flow in the Sitting Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lashmi Venkatraghavan (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor-Investigator, Lashmi Venkatraghavan, Assistant Professor, Department of Anesthesia, Toronto Western Hospital, Toronto, Canada, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-8319
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Jugular Venous Flow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sitting position (Experimental): The volunteers were kept comfortable in the sitting position. The cricoid cartilage (representing the C6 level) was used as a landmark. A horizontal straight line drawn across the volunteer's neck at the cricoid level and intersecting the IJV on both sides of the neck marked the initial scanning points. The second scanning point was along the IJV at the highest accessible point on the neck. Internal jugular vein cross-sectional area and blood velocity were measured using 2D ultrasound and Doppler (Philips CX50, Andover, MA, USA), respectively, with a 12-3 MHz transducer (Philips L12-3, Andover, MA, USA)
  Interventions: Diagnostic Test: Jugular venous ultrasound

INTERVENTIONS:
Diagnostic Test: Jugular venous ultrasound — All volunteers will be fully awake throughout the study and be kept comfortable. A cross will be marked where the left and right IJV cross the level of C6. This is where all the measurements will be taken in 3 different conditions at rest, jugular occlusion and valsalva maneuver. At each conditions, the left and right IJV will be scanned with an ultrasound measuring the cross sectional area and Doppler velocity of the IJV. The least amount of pressure will be used to press on the ultrasound probe and the measurements will be obtained at end inspiration. The IJV flow is then calculated.

SUMMARY:
During neurosurgical procedures, patients need to be placed in sitting position for surgical access especially in surgeries in the vertex or posterior fossa. Due gravitational effect of sitting position the flow in IJV may be reduced. Venous air embolism (VAE) is a common complication of sitting position craniotomy and carries high mortality and morbidity. Venous pressure decreases as the head of the patient is raised above the heart. Hence, negative venous pressure in the cerebral venous system promotes entrapment of air in accidental opening of the sinuses.

Common methods to prevent VAE in sitting position include increasing the venous pressure by either jugular venous compression and/or increasing the venous pressure by adding positive end expiratory pressure (PEEP). Both these methods can decrease venous return and can lead to brain swelling.. In addition, improper neck position can cause the kinking of the IJV which may lead to decreased venous drainage and increased ICP. This has been shown to be the contributing factor for intraoperative brain swelling and postoperative neck and tongue swelling leading to airway obstruction. Optimal brain perfusion is best in the neutral position of the head, but surgery cannot always be performed with this.

DETAILED DESCRIPTION:
Currently, there are no studies that looked into the IJV flow in sitting position and effect of venous outflow obstruction on the IJV flow. Valsalva maneuver (forced inspiration with closed glottis) and /or compression of internal jugular veins (IJV) are the two commonly used physiological methods that can cause venous outflow obstruction. A custom made neck collar can be used for compression of internal jugular vein and previous investigations have used a similar device in a rat model to demonstrate the protective effects on slosh-mediated brain injury by increasing intracranial blood volume . While the collars have not yet been studied on people for their effectiveness at preventing concussions, many studies have looked at the effect of neck collars on both jugular compression and ICP..

The purpose of this study is to measure the venous blood flow of healthy volunteers by the use of an ultrasound and Doppler velocimetry in sitting position. the investigators will measure the IJV flow on both sides in sitting position at rest and at two conditions of venous outflow obstruction- 1. Neck compression using a custom made collar and 2. During 30 seconds Valsalva maneuver. This study will provide information on the cerebral venous drainage. This information will be very useful in planning and positioning of patients undergoing neurosurgical procedures and to prevent complications from the improper patient position.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers who are above the age of 18 ASA 1
* Body mass index (BMI) less than and equal to 35

Exclusion Criteria:

* Lack of informed consent
* Language barrier
* Medical students and anesthesia residents going through the department as part of their rotation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lashmi Venkatraghavan, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Internal Jugular Vein Flow in the Sitting Position: The volunteers were kept comfortable in the sitting position. The cricoid cartilage (representing the C6 level) was used as a landmark. A horizontal straight line drawn across the volunteer's neck at the cricoid level and intersecting the IJV on both sides of the neck marked the initial scanning points
Period: Overall Study
Arm/Group | Internal Jugular Vein Flow in the Sitting Position
Started | 12
Completed | 10
Not Completed | 2
Not completed — poor compliance | 2

BASELINE CHARACTERISTICS:
Population: Data analyzed for only 10 participants who completed the study, two participants were excluded from the study due to poor compliance.
Groups:
- Sitting Position: The volunteers were kept comfortable in the sitting position. The cricoid cartilage (representing the C6 level) was used as a landmark. A horizontal straight line drawn across the volunteer's neck at the cricoid level and intersecting the IJV on both sides of the neck marked the initial scanning points
Arm/Group | Sitting Position
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants] — Population: Out of 12 participants, 10 participants completed the study, two participants were excluded from the study due to poor compliance.
  Participants
    healthy adult volunteers>18 yr: number analyzed (Participants) | 10
    healthy adult volunteers>18 yr: <=18 years | 0
    healthy adult volunteers>18 yr: Between 18 and 65 years | 10
    healthy adult volunteers>18 yr: >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Out of 12 participants, 10 participants completed the study, two participants were excluded from the study due to poor compliance.
  Participants
    number analyzed (Participants) | 10
    Female | 2
    Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Internal Jugular Venous Flow
Description: Right Internal Jugular Vein Flow in the sitting position.
Time Frame: 1 day
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: cm2
Groups:
- Right IJV at Rest: Venous Jugular Flow in the Sitting Position at rest on right Internal Jugular Venous
- Right IJV With Collar: Venous Jugular Flow in the Sitting Position with collar on right Internal Jugular Venous
Arm/Group | Right IJV at Rest | Right IJV With Collar
Number analyzed (Participants) | 10 | 10
cm2
  Cross-sectional area at C6 | 0.04 [0.03 to 0.08] | 0.4 [0.2 to 0.6]
  High cross-sectional area | 0.04 [0.02 to 0.06] | 0.21 [0.17 to 0.30]

2. Primary Outcome: Left Internal Jugular Vein Flow
Description: left internal jugular vein cross-sectional area in the sitting position at rest and with application of the cervical collar.
Time Frame: 1 day
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: cm2
Groups:
- Left IJV at Rest: Venous Jugular Flow in the Sitting Position at rest on left Internal Jugular Venous
- Left IJV With Collar: Venous Jugular Flow in the Sitting Position with collar on left Internal Jugular Venous
Arm/Group | Left IJV at Rest | Left IJV With Collar
Number analyzed (Participants) | 10 | 10
cm2
  Cross-sectional area at C6 | 0.07 [0.05 to 0.13] | 0.35 [0.17 to 0.44]
  High cross-sectional area | 0.05 [0.03 to 0.09] | 0.13 [0.11 to 0.15]

3. Primary Outcome: Right Internal Jugular Vein Flow in the Sitting Position
Description: Right internal jugular vein peak velocity in the sitting position at rest and with application of the cervical collar
Time Frame: one day
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: cm.sec-1
Groups:
- Right Internal Jugular Vein in the Sitting Position at Rest; Right Internal Jugular Vein in the Sitting Position Collar: The volunteers were kept comfortable in the sitting position. The cricoid cartilage (representing the C6 level) was used as a landmark. A horizontal straight line drawn across the volunteer's neck at the cricoid level and intersecting the IJV on both sides of the neck marked the initial scanning points
Arm/Group | Right Internal Jugular Vein in the Sitting Position at Rest | Right Internal Jugular Vein in the Sitting Position Collar
Number analyzed (Participants) | 12 | 12
cm.sec-1 | 70 [9 to 116] | 17 [10 to 22]

4. Primary Outcome: Right Internal Jugular
Description: Comparisons of right internal jugular vein ﬂow in the sitting position at rest and with application of the cervical collar
Time Frame: one day
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: mL.min-1
Groups:
- Right Internal Jugular Vein in the Sitting Position Collar: Comparisons of bilateral internal jugular vein cross-sectional area, peak velocity, and ﬂow in the sitting position at rest and with application of the cervical collar
Arm/Group | Right Internal Jugular Vein in the Sitting Position at Rest | Right Internal Jugular Vein in the Sitting Position Collar
Number analyzed (Participants) | 10 | 10
mL.min-1
  Flow at C6 | 193 [50 to 491] | 349 [262 to 488]
  Flow at high cross-sectional area | 121 [23 to 328] | 236 [114 to 503]

5. Secondary Outcome: Left Internal Jugular Vein Flow in the Sitting Position
Description: Comparisons of left internal jugular vein peak velocity in the sitting position at rest and with application of the cervical collar
Time Frame: One day
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: cm.sec-1
Arm/Group | Left IJV at Rest | Left IJV With Collar
Number analyzed (Participants) | 10 | 10
cm.sec-1 | 30 [22 to 47] | 12 [5 to 16]

6. Secondary Outcome: Left Internal ﬂow in the Sitting Position
Description: left internal jugular vein ﬂow in the sitting position at rest and with application of the cervical collar
Time Frame: One day
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: mL.min-1
Arm/Group | Left IJV at Rest | Left IJV With Collar
Number analyzed (Participants) | 10 | 10
mL.min-1
  Flow at C6 | 113 [93 to 323] | 183 [78 to 389]
  Flow at high cross-sectional area | 105 [38 to 170] | 889 [36 to 1742]

ADVERSE EVENTS:
Time Frame: 1 day
Description: Any adverse events detected during the procedure
Groups:
- Internal Jugular Venous Flow in Sitting Position: The volunteers were kept comfortable in the sitting position. The cricoid cartilage (representing the C6 level) was used as a landmark. A horizontal straight line drawn across the volunteer's neck at the cricoid level and intersecting the IJV on both sides of the neck marked the initial scanning points
Arm/Group | Internal Jugular Venous Flow in Sitting Position
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes